CLINICAL TRIAL: NCT00177190
Title: In Vitro Evaluation of Immune Responses in CTCL
Brief Title: In Vitro Evaluation of Immune Responses in Cutaneous T-Cell Lymphoma (CTCL)
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Larisa Geskin, Associate Professor of Dermatology, University of Pittsburgh
Other Study IDs: 0307015
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2013-06

CONDITIONS: Cutaneous T-cell Lymphoma; Sezary Syndrome; Mycosis Fungoides
Keywords: Cutaneous T-cell Lymphoma; Sezary Syndrome; Mycosis Fungoides; Immune Responses
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Sezary Syndrome; Mycosis Fungoides

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — White cells
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is an in vitro evaluation of cutaneous T-cell lymphoma using patients' blood and tissue to evaluate immune responses related to identified tumor populations and dendritic/CD 8 cells.

DETAILED DESCRIPTION:
This is an in vitro evaluation of cutaneous T-cell lymphoma using patients blood and tissue to evaluate immune responses related to identified tumor populations and dendritic/ CD 8 cells with the following objectives:

* Objective I: Evaluate the feasibility of the preparation of dendritic cells (DCs), CD8 and Sezary cells (all CD4 positive) in vitro, obtained from the buffy coats or a skin biopsy from an area with tumor involvement of subjects with cutaneous t-cell lymphoma (CTCL) and Sezary syndrome (leukemic stage of CTCL) undergoing an approved FDA therapy, extracorporeal photopheresis (ECP).
* Objective II: Evaluate antigen loading of the DCs.
* Objective III: Test the functional capacities of the DCs derived from CTCL subjects to overcome immune tolerance to the tumor cells ex-vivo, by using modified Elispot assay in conjunction with Granzyme B Elispot assay as a measurement of cytotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Males or females <18 years of age
* Histologically confirmed stage IV cutaneous T-cell lymphoma, with at least 5% of the peripheral blood lymphocytes showing atypical morphology consistent with Sezary cells
* Ambulatory and be in stable medical condition
* Biopsy positive mycosis fungoides/CTCL or clonal type of CTCL as determined by PCR for TCR and Southern blot for TCR

Exclusion Criteria:

* Received any chemotherapy or radiotherapy within 4 weeks prior to enrollment
* Significant psychiatric illness which would prevent adequate informed consent in the opinion of the principal investigator
* Systemic steroid therapy other than maintenance for adrenal suppression
* Known coagulopathy for non SS subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cutaneous Lymphoma Clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2002-06; Primary Completion 2005-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Functional capacity of dendritic cells in-vitro | At each cell collection
  Evaluate the feasibility of the preparation of dendritic cells (DCs), CD8 and Sezary cells (all CD4 positive) in vitro, obtained from the buffy coats or a skin biopsy from an area with tumor involvement of subjects with cutaneous t-cell lymphoma (CTCL) and Sezary syndrome (leukemic stage of CTCL)

SECONDARY OUTCOMES:
Evaluate antigen loading of dendritic cells | At each cell collection
  Functional DCs can be isolated and effectively loaded with the malignant cells by several methods (coculture and fusion)

CONTACTS AND LOCATIONS:
Overall Officials: Larisa J. Geskin, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States